CLINICAL TRIAL: NCT00794131
Title: Phase I Study of the Safety, Tolerability,and Tumor-Specific Replication of the Intravenous Administration of Green Fluorescent Protein Encoded Genetically Engineered Attenuated Vaccinia Virus, GL-ONC1, in Patients With Advanced Solid Organ Cancers.
Brief Title: Safety Study of GL-ONC1, an Oncolytic Virus, in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genelux GmbH (Industry)
Responsible Party: Sponsor
Organization: Genelux Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL-ONC1-002/MA
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Advanced Cancers (Solid Tumors)
Keywords: cancer; vaccinia virus; vaccinia; oncolytic; oncolytic virus; biological; imaging
MeSH Terms: conditions — Neoplasms; Vaccinia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: GL-ONC1 — a genetically-engineered vaccinia virus (encoding Renilla luciferase-Aequorea green fluorescent protein fusion, β-galactosidase, and β-glucuronidase )

SUMMARY:
The main purpose of this study is to determine whether, GL-ONC1, an Oncolytic Virus, can safely be administered intravenously in patients with advanced solid tumors.

DETAILED DESCRIPTION:
In preclinical studies, GL-ONC1 an oncolytic vaccinia virus, has shown the ability to preferentially locate, colonize and destroy tumor cells. This study seeks to evaluate the safety profile of an attenuated vaccinia virus when administered intravenously to patients with advanced solid tumors. The study also seeks to detect virus delivery to primary and/or metastatic tumors, including evaluation of viral delivery by fluorescence imaging (GFP expression); whether anti-vaccinia virus immune response occurs; and will record evidence of any anti-tumor activity. For Cohorts 8 and Expansion Cohort 1B, CTC counts, virus-encoded marker gene analysis and Dynamic Contrast (DCE-MRI) MRI imaging will be used to evaluate tumor micro-circulation in vivo. These measures will be evaluated for their potential predictive value of survival outcomes, and to evaluate any correlation of such pharmacodynamic and response rate indicators in the GL-ONC1 treatment context.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically documented, advanced stage, primary or metastatic solid tumors refractory to standard therapy or for which no curative standard therapy exists.
* Evidence of measurable or evaluable disease.
* Age must be ≥ 18 years.
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedures must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, Version 3.0) Grade ≤ 1. Surgery must have occurred at least 28 days prior to study enrolment.
* Chemotherapy or radiotherapy (other than small-field palliative radiotherapy), immunotherapy and/or hormonal therapy must have been received > 28 days prior to receiving study drug. Subjects may continue to receive LHRH analogue therapy for prostate cancer in face of rising PSA. Bisphosphonates and anticoagulants are permitted.
* ECOG Performance Score ≤ 1.
* Life expectancy of at least 3 months.
* Required baseline laboratory data include:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9 [SI units 10^9/L]
  * Platelets ≥ 100 x 10^9 [SI units 10^9/L]
  * Haemoglobin ≥ 9.0 g/dL [SI units gm/L]
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Bilirubin ≤ 1.5 x ULN
  * AST/ALT ≤ 2.5 x ULN or ≤ 5 x ULN in the presence of liver metastases
* Ejection fraction of ≥50% by MUGA or ECHO.
* Signed informed consent indicating that the subject is aware of the neoplastic nature of his or her disease and has been informed of the procedures to be followed, the experimental nature of the therapy, the alternatives and the potential benefits, side effects, risks, and discomforts.
* Willing and able to comply with scheduled visits, treatment plan, and laboratory tests.
* Female patients must have a negative pregnancy test within five days prior to treatment.
* Female patients of childbearing potential who are not surgically sterile or postmenopausal and male patients who are not surgically sterile must agree to use highly effective contraception. Barrier methods for contraception must be applied during the treatment period and up to day 60 after the last virus application. The patient must agree to sign his or her consent on this particular inclusion criterion.

Additional Inclusion Criteria Relevant for Cohort 8 and the Phase IB Expansion Cohort:

1. Diagnosis of histologically or cytologically documented, advanced stage solid tumor (e.g., primary or metastatic breast, prostate or colorectal cancer) refractory to standard therapy or for which no curative standard therapy exists.
2. Evidence of measurable or evaluable disease.
3. Disease that can be safely serially biopsied.
4. Circulating tumor cell count > 10 for analyses of tumor cell viral delivery.

Exclusion Criteria:

* Prior therapy with a cytolytic virus of any type.
* Concurrent therapy with any other investigational anticancer agent.
* Concurrent vaccines or immunotherapy during, and for 30 days before or after, study therapy.
* Concurrent antiviral agent active against vaccinia virus (e.g. cidofovir, vaccinia immunoglobulin, imatinib, ST-246) during course of study.
* Patients vaccinated with vaccinia virus within the past 10 years.
* Patients with known brain metastases: due to poor prognosis and risk of developing progressive neurological dysfunction that would confound the evaluation of neurological or other adverse events.
* Patients with known allergy to ovalbumin or other egg products.
* Patients with immune system disorders or who are receiving immunosuppressive therapy or any steroids.
* Patients with clinically significant dermatological disorders, e.g. eczema or psoriasis, or any unhealed skin wounds or ulcers, as assessed by the principal investigator during the screening and during the study.
* Patients with fevers, or any systemic infections, including known HIV infection, hepatitis B or C.
* Prior splenectomy.
* Previous organ transplant.
* Pregnant or breast-feeding women.
* Clinically significant cardiac disease (New York Heart Association, Class III or IV) including pre-existing arrhythmia, uncontrolled angina pectoris or myocardial infarction within one year prior to study entry, or grade 2 or higher compromised left ventricular ejection fraction (as determined by MUGA).
* Dementia or altered mental status that would prohibit informed consent.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the principal investigator, would make the subject inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of GL-ONC1, administered intravenously to patients with advanced solid tumors. | Every 30 minutes for 2 hours after each administration of GL-ONC1, then daily until discharge and on day 8, then weekly up to day 21, then week 12 and week 24

SECONDARY OUTCOMES:
Detection of virus delivery to primary and/or metastatic tumors by PCR and immunohistochemistry. | To be performed where tumor is deemed safely accessible for biopsy (requires patient consent). Timing of post-treatment biopsy may vary to optimise data generated, however, within two weeks of administration is considered suitable.
Evaluation of anti-vaccinia virus immune response (antibody responses) | To be done at baseline and weekly for the first 8 weeks for all cohorts. A final test will be performed on day 30 after the last virus application.
Evaluation of viral delivery by fluorescence imaging | The timing and frequency of visualization will be dependent on the acquired data but may be pursued once weekly for the length of the observation period.
Determine recommended dose and schedule for future investigation. | At the end of the study
Evaluation of anti-tumor activity | Week 12 and week 24 after each cycle (Cohorts 1-7). Cohort 8, 1B: 15 days (± 3 days),on D 29 (± 3 days) prior to Cycle 2 ;CT: weeks 12, 24
  Generally CT scan (conventional or spiral), PET/CT, MRI or clinical examination will be used for patients in Cohorts 1-7, however tumor markers can also be used to assess response. For patients enrolled in Cohort 8 and the Phase IB expansion cohort of this trial, tumor evaluation will also be performed by DCE and DW-MRIs as well as FDG-PET-CT and CT scans. RECIST and modified CHOI criteria for response will be employed in image evaluations.
Determine possible predictive value of Circulating Tumor Cell counts and Beta-glucuronidase levels relative to patient survival outcomes. | CTC's: baseline, Cycle 1 Day 8, prior to dosing D 1 of Cycles 2, 3, 4. Beta-glucuronidase analysis: baseline , weekly first 2 cycles, monthly pre-dose for following cycles;.Final test day 30 after last treatment
  Circulating Tumor Cells are present in patients with advanced metastatic solid tumor cancers. Beta-glucomidase analysis will be used to determine expression of the virus encoded marker genes. CTC counts and Beta-glucomidase values together may be a prognostic indicator (measure of survival outcomes) for patients with solid tumors.
Assess correlation of CTC number with radiological (imaging) as early pharmacodynamic and response rate indicators for GL-ONC1 treatment. | CTC's: baseline, Cycle 1 Day 8, prior to dosing Day 1 of Cycles 2, 3, 4. Imaging: DCE, DW-MRIs and FDG-PET-CT at baseline, 15 days, on Day 29 prior to administration of Cycle 2; CT scans: weeks 12,24.
  For patients in Cohort 8 and a Phase 1B expansion study group who have high circulating blood cell counts and solid tumors that may be safely, serially biopsied, the study seeks to demonstrate the correlation of CTC number with radiological outcomes, including Dynamic Contrast Enhanced (DCE) and Diffusion Weighted (DW) magnetic resonance imaging (MRI) and fluoro-deoxy glucose (FDG)-positron emission tomography (PET)-computed tomography (CT) scan changes as early pharmacodynamic and response rate indicators in the GL-ONC1 treatment context.

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, MD FRCP MSc PhD, Principal Investigator — Royal Marsdon Hospital/Institute for Cancer Research; Kevin Harrington, MBBS MRCP FRCR, Principal Investigator — Royal Marsden Hospital/Institute of Cancer Research; Hardev Pandha, MD,FRCP,FRACP,PhD, Principal Investigator — Surrey Clinical Research Centre
Locations (1):
- Royal Marsden Hospital, Surrey, United Kingdom

REFERENCES:
- See also: Click Here for more information about this study: Safety Study of GL-ONC1, an Oncolytic Virus, in Patients with Advanced Solid Tumors — http://www.genelux.com